CLINICAL TRIAL: NCT05300204
Title: Evaluating the Efficacy and the Acceptability of the Website "Ich Bin Alles" to Improve Depression Literacy in Adolescents With Acute or Remitted Major Depressive Disorder
Brief Title: Evaluation of a Website to Improve Depression Literacy in Adolescents With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Prof. Otto Beisheim Foundation (Other)
Responsible Party: Principal Investigator, Ellen Greimel, Postdoctoral Researcher, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20114_2
Record Dates: First submitted 2022-03-10; First posted 2022-03-29 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Depressive Disorder; Depression in Adolescence
Keywords: Knowledge; Mental Health; Depression Literacy; Website; Online; Adolescence; Youth
MeSH Terms: conditions — Depressive Disorder; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two intervention groups in parallel for the duration of the study
Who Masked: Participant
Masking Description: Participants are not aware of the assigned intervention group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group 1 - Self-help Strategies for depression (Experimental): Exposure to information about self-help strategies for depression
  Interventions: Other: Self-help strategies for depression
- Intervention Group 2 - General information about depression (Experimental): Exposure to general information about depression
  Interventions: Other: General information about depression

INTERVENTIONS:
Other: Self-help strategies for depression — Before starting the intervention, the participants are told that they will be shown parts of a website about depression. The participants are instructed to carefully attend to the website (e.g., to read the text precisely, to hear attentively to the podcasts and to view carefully the videos and images on the website). The time window spent for the reception of each part of the website are fixed.
  The participants in this intervention group will only be shown parts of the website regarding self-help strategies for depression.
  Arms: Intervention Group 1 - Self-help Strategies for depression
Other: General information about depression — Before starting the intervention, the participants are told that they will be shown parts of a website about depression. The participants are instructed to carefully attend to the website (e.g., to read the text precisely, to hear attentively to the podcasts and to view carefully the videos and images on the website). The time window spent for the reception of each part of the website are fixed.
  The participants in this intervention group will only be shown parts of the website regarding general information about depression
  Arms: Intervention Group 2 - General information about depression

SUMMARY:
The aim of this study is to evaluate the efficacy and acceptability of the website "ich bin alles" (https://www.ich-bin-alles.de/) to improve depression literacy (knowledge about depression, which aid the recognition, treatment or prevention of depression) in adolescents with acute or remitted depressive disorder. The investigators will examine whether the website improves depression literacy in adolescents aged 12 to 18 years with a history of depression. The investigators will also assess the acceptability of the website among the adolescents.

DETAILED DESCRIPTION:
Few young people with major depressive disorder seek professional treatment in time. Concerns about social stigma, confidentiality, and limited knowledge about mental health conditions, such as depression, or mental health services are some of the main barriers to seek treatment. To address these problems, we developed an evidence-based website "ich bin alles" (https://www.ich-bin-alles.de/) to improve depression literacy.

To improve depression literacy, the website provides general information about depression as psychiatric disorder in adolescents (e.g., symptoms, causes, course and treatment of depression). Furthermore, the website provides information about self-help strategies for depression and prevention of depression; i.e., strategies for promoting mental health (e.g., reducing stress, doing exercise, undertaking positive activities), which are meant to serve as an addition to professional treatments of depression or to promote mental health in adolescents.

Target groups of the website are adolescents aged 12 to 18 years seeking help for depression, as well as healthy adolescents seeking information about mental health promotion or depression. Easy access to information about depression would make early recognition of depression more likely and engage young people to seek help for depression.

Since the website targets two different groups, the investigators will evaluate the website accordingly:

Target group 1: Adolescents with a major depressive disorder (acute or remitted) Target group 2: Healthy Adolescents (no mental health condition)

The current study will focus on target group 1. A study focusing on target group 2 can be found in a separately registered clinical trial on clinicaltrials.gov.

The primary aim of this study is to evaluate the efficacy and acceptability of the website "ich bin alles" (https://www.ich-bin-alles.de/) to improve depression literacy in adolescents with acute or remitted depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* The presence of a current or remitted diagnosis of a mild, moderate, or severe major depressive episode according to ICD-10 Criteria: F32.0; F32.1; F32.2, F33.0, F33.1, F.33.2) is assessed using a semi structured clinical Interview: the "Kinder-DIPS". The Kinder-DIPS is a well-established German interview for the diagnosis of a wide range of axis I psychiatric disorders in children from ages six to 18.
* Depressive symptomatology is measured as well with the Beck Depression Inventory Second Edition (BDI-II) for descriptive purposes. The BDI-II is a self-report inventory to assess the severity of depressive symptoms, rated on a 4-point response scale, with higher scores indicating more severe depressive symptoms.
* Intelligence quotient (IQ) of ≥ 80.

Exclusion Criteria:

* Acute suicidality
* Schizophrenic disorder
* Pervasive developmental disorder
* Bipolar disorder
* Borderline personality disorder
* Substance dependence disorder
* Insufficient knowledge of German

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Depression Literacy - Self-help Strategies | Pre-Test, Post-Test (within 2 hours), Follow-Up 1 (Week 2), Follow-Up 2 (Week 4)
  This self-designed questionnaire is a self-report inventory to assess knowledge of self-help strategies for depression (12 items), with higher scores indicating more knowledge of self-help strategies. Participants will complete this self-designed questionnaire at pre-test, post-test and the two follow-ups to determine change in knowledge of self-help strategies.
Depression Literacy - Depression as psychiatric disorder | Pre-Test, Post-Test (within 2 hours), Follow-Up 1 (Week 2), Follow-Up 2 (Week 4)
  This self-designed questionnaire is a self-report inventory to assess knowledge of depression as psychiatric disorder (frequency and comorbidities, treatment, symptoms, causes and course of depression; 27 items), with higher scores indicating more knowledge of depression as psychiatric disorder. Participants will complete this self-designed questionnaire at pre-test, post-test and the two follow-ups to determine change in knowledge of depression as psychiatric disorder

SECONDARY OUTCOMES:
Visual Aesthetics of Websites Inventory Short Version (VisAWI-S) | Post-Test (within 2 hours)
  The short version of the Visual Aesthetics of Websites Inventory (VisAWI-S) is self-report inventory to assess the evaluation of the website's design - especially the perceived visual aesthetics. Participants indicated their response to the four items (e.g., "The layout appears professionally designed") on a seven-point Likert scale (ranging from 1 "do not agree at all" to 7 "do fully agree")
Overall reception of the website | Post-Test (within 2 hours)
  The overall reception of the website as measured with a self-designed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Schulte-Körne, Professor, Study Director — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University Hospital Munich
Locations (1):
- Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University Hospital Munich, Munich, Germany, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Data in our study contains sensitive patient information, such as sociodemographic information and comorbidities. Since patients could possibly be identified by making our raw data publicly available, ethical principles of protecting patient confidentiality would be breached. Aggregated group data can be made available upon request.

REFERENCES:
- [Derived] Kloek MWH, Primbs R, Kaubisch S, Iglhaut L, Piechaczek CE, Zsigo C, Keim PM, Feldmann L, Schulte-Korne G, Greimel E. Effectiveness and acceptance of tailored web-based psychoeducation for adolescents with major depression. Patient Educ Couns. 2026 Feb;143:109429. doi: 10.1016/j.pec.2025.109429. Epub 2025 Nov 27. PMID 41337834